CLINICAL TRIAL: NCT06439615
Title: The Treatment Effect of Baricitinib for the Secondary Pulmonary Complications Following Spontaneous Subarachnoid Hemorrhage
Brief Title: Baricitinib for the Lung Injury Following Spontaneous SAH
Acronym: BLISS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BAR-SAH
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Spontaneous Subarachnoid Hemorrhage
Keywords: Spontaneous subarachnoid hemorrhage; Baricitinib; Inflammation; Complications; Acute respiratory distress syndrome; Pneumonia; Outcome
MeSH Terms: conditions — Subarachnoid Hemorrhage; Inflammation; Respiratory Distress Syndrome; Pneumonia | interventions — baricitinib; Janus Kinase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control group (Sham Comparator): Participants will receive standard treatment and care according to the current management guidelines for SAH.
  Interventions: Other: Standard treatment
- Baricitinib group (Experimental): In addition to receiving standard treatment and care, baricitinib will be administrated orally (or crushed for nasogastric tube delivery) at a daily dosage of 4mg for three consecutive days following SAH.
  Interventions: Drug: Baricitinib 4 MG; Other: Standard treatment

INTERVENTIONS:
Drug: Baricitinib 4 MG — Baricitinib will be administered orally (or crushed for nasogastric tube delivery) at a daily dosage of 4mg for three consecutive days following SAH.
  Other Names: JAK Inhibitor
  Arms: Baricitinib group
Other: Standard treatment — Participants will receive standard treatment and care according to the current management guidelines for subarachnoid hemorrhage.

SUMMARY:
The present study is a randomized, parallel control, and double-blind trial designed to assess the efficacy of baricitinib in reducing the occurrence of pulmonary complications in patients with spontaneous subarachnoid hemorrhage (SAH). The research protocol incorporates an adaptive design, allowing for modifications to key elements such as the sample size enrolled during interim analysis.

DETAILED DESCRIPTION:
Subarachnoid hemorrhage (SAH) is an acute cerebrovascular disorder resulting from the rupture of intracranial vessels, primarily caused by factors such as the rupture of intracranial aneurysms (accounting for approximately 75%-80% of SAH cases), arteriovenous malformations, and abnormal vasculature.

Pulmonary complications, including pneumonia and acute respiratory distress syndrome (ARDS), frequently manifest in a significant number of subarachnoid hemorrhage (SAH) patients, significantly impacting their prognosis. The pathogenesis of these complications can be partially attributed to an exaggerated inflammatory response during the acute phase following SAH. The incidence of cerebrovascular spasm and mortality rates significantly increase in SAH patients with pulmonary complications, thereby resulting in a poorer long-term prognosis. However, the current strategy for preventing or managing pulmonary complications after SAH is not sufficiently effective.

The JAK-STAT signaling pathway, a pivotal stress-induced inflammatory cascade triggered subsequent to SAH, is characterized by its rapid response to external stimuli. Baricitinib, a JAK inhibitor developed by Eli Lilly Company, exerts significant anti-inflammatory effects in diverse pathological processes and finds extensive application in patients with rheumatoid arthritis, COVID-19, and alopecia areata. However, it remains uncertain whether early administration of baricitinib can mitigate the incidence of secondary pulmonary complications and enhance the prognosis of SAH by suppressing the exaggerated inflammatory response during the acute phase following SAH.

The current multicenter clinical trial is designed as a randomized, parallel control, and double-blind study to assess the efficacy of baricitinib in reducing pulmonary complications among patients with SAH. SAH Patients admitted to participating clinical centers with a Hunt-Hess score of Ⅲ-Ⅳ will undergo continuous screening based on predefined selection criteria. The enrolled subjects will be randomly allocated into an experimental group and a control group, receiving either Baricitinib (4mg/day for 3 days) in addition to conventional treatment or placebo in addition to conventional treatment, respectively. The primary outcome is the incidence of pneumonia within 14 days after SAH. While the secondary outcome including the incidence of ARDS and other pulmonary complications within 14 days, the incidence of serious adverse events within 14 days, the proportion of patients requiring assisted ventilation measures within 14 days, the mortality rate within 14/30/90 days, as well as the neurological outcome at 30/90 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤80 years old;
2. Diagnosed with spontaneous subarachnoid hemorrhage through imaging or lumbar puncture;
3. Hunt-Hess score of Ⅲ-Ⅳ;
4. Acute onset, admitted to the hospital within 24 hours of onset

Exclusion Criteria:

1. Presence of lung diseases before initiation of study treatment such as chronic obstructive emphysema, bronchiectasis, lung cancer, tuberculosis, or a history of lung surgery;
2. Presence of autoimmune diseases, immune system dysfunction, or blood system dysfunction (absolute lymphocyte count (ALC) less than 0.5×109 cells/L, absolute neutrophil count (ANC) less than 1×109 cells/L, or hemoglobin value less than 8 g/dL) before the onset of the disease;
3. Secondary SAH (such as traumatic SAH), or combined craniocerebral trauma, intraparenchymal hemorrhage, or peripheral organ trauma;
4. Evidence of fever or infection already present at the time of admission;
5. History of previous craniocerebral surgery, previous cerebral hemorrhage, craniocerebral injury, cerebral infarction, intracranial tumor, or presence of neurological dysfunction before the onset of the disease;
6. Presence of contraindications for baricitinib treatment, including severe liver damage, renal dysfunction (creatinine clearance rate <30ml/min), hypercholesterolemia, or known drug allergies;
7. Taking JAK inhibitors or other immunosuppressive drugs before the onset of the disease;
8. Expected survival time less than 2 weeks;
9. Females who are pregnant or breastfeeding;
10. Currently participating in other interventional clinical studies;
11. Patients who refuse to sign the consent form or refuse to accept follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of pneumonia | up to 14 days
  Proportion of patients who occur pneumonia within 14 days

SECONDARY OUTCOMES:
The incidence of ARDS | up to 14 days
  The incidence of ARDS within 14 days following SAH.
The incidence of other pulmonary complications | up to 14 days
  The incidence of additional pulmonary complications, such as pulmonary edema, pulmonary embolism, and pleural effusion among patients within 14 days following SAH.
The incidence of assisted ventilation measures | up to 14 days
  The proportion of patients requiring assisted ventilation measures within 14 days following SAH.
The incidence of Systemic Inflammatory Response Syndrome(SIRS) | up to 14 days
  The incidence of SIRS within 14 days following SAH.
Mortality rate | up to 90 days
  The mortality rate within 14 days / 30 days / 90 days.
The incidence of serious adverse events (SAE) | up to 14 days
  The incidence of SAE within 14 days following SAH.
The neurological functional outcome | up to 90 days
  The neurological functional scores evaluated by Modified Rankin Scale and Glasgow Outcome Scale at 30 days and 90 days after SAH.
The cognitive impairment after SAH | up to 90 days
  The Mini-Mental Status Exam (MMSE) scores at 90 days after SAH.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Qu, PhD MD, Principal Investigator — Department of Neurosurgery, Tangdu Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robba C, Busl KM, Claassen J, Diringer MN, Helbok R, Park S, Rabinstein A, Treggiari M, Vergouwen MDI, Citerio G. Contemporary management of aneurysmal subarachnoid haemorrhage. An update for the intensivist. Intensive Care Med. 2024 May;50(5):646-664. doi: 10.1007/s00134-024-07387-7. Epub 2024 Apr 10. PMID 38598130
- [Background] Chai CZ, Ho UC, Kuo LT. Systemic Inflammation after Aneurysmal Subarachnoid Hemorrhage. Int J Mol Sci. 2023 Jun 30;24(13):10943. doi: 10.3390/ijms241310943. PMID 37446118
- [Background] Kahn JM, Caldwell EC, Deem S, Newell DW, Heckbert SR, Rubenfeld GD. Acute lung injury in patients with subarachnoid hemorrhage: incidence, risk factors, and outcome. Crit Care Med. 2006 Jan;34(1):196-202. doi: 10.1097/01.ccm.0000194540.44020.8e. PMID 16374174
- [Background] Macmillan CS, Grant IS, Andrews PJ. Pulmonary and cardiac sequelae of subarachnoid haemorrhage: time for active management? Intensive Care Med. 2002 Aug;28(8):1012-23. doi: 10.1007/s00134-002-1382-7. Epub 2002 Jul 6. PMID 12185419
- [Background] RECOVERY Collaborative Group. Baricitinib in patients admitted to hospital with COVID-19 (RECOVERY): a randomised, controlled, open-label, platform trial and updated meta-analysis. Lancet. 2022 Jul 30;400(10349):359-368. doi: 10.1016/S0140-6736(22)01109-6. PMID 35908569
- [Background] Taylor PC, Laedermann C, Alten R, Feist E, Choy E, Haladyj E, De La Torre I, Richette P, Finckh A, Tanaka Y. A JAK Inhibitor for Treatment of Rheumatoid Arthritis: The Baricitinib Experience. J Clin Med. 2023 Jul 6;12(13):4527. doi: 10.3390/jcm12134527. PMID 37445562
- [Background] Ely EW, Ramanan AV, Kartman CE, de Bono S, Liao R, Piruzeli MLB, Goldman JD, Saraiva JFK, Chakladar S, Marconi VC; COV-BARRIER Study Group. Efficacy and safety of baricitinib plus standard of care for the treatment of critically ill hospitalised adults with COVID-19 on invasive mechanical ventilation or extracorporeal membrane oxygenation: an exploratory, randomised, placebo-controlled trial. Lancet Respir Med. 2022 Apr;10(4):327-336. doi: 10.1016/S2213-2600(22)00006-6. Epub 2022 Feb 3. PMID 35123660
- [Background] Taylor PC, Keystone EC, van der Heijde D, Weinblatt ME, Del Carmen Morales L, Reyes Gonzaga J, Yakushin S, Ishii T, Emoto K, Beattie S, Arora V, Gaich C, Rooney T, Schlichting D, Macias WL, de Bono S, Tanaka Y. Baricitinib versus Placebo or Adalimumab in Rheumatoid Arthritis. N Engl J Med. 2017 Feb 16;376(7):652-662. doi: 10.1056/NEJMoa1608345. PMID 28199814